CLINICAL TRIAL: NCT03532282
Title: Randomized Controlled Study of the Effectiveness of Stepped-Care Sleep Therapy In General Practice
Brief Title: The RESTING Insomnia Study: Randomized Controlled Study on Effectiveness of Stepped-Care Sleep Therapy
Acronym: RESTING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rachel Manber, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 45874; R01AG057500 (NIH)
Record Dates: First submitted 2018-05-01; First posted 2018-05-22 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are asked to refrain from mentioning any information about the treatment they receive when interacting with the investigator or outcomes assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONLINE ONLY (Active Comparator): Online cognitive behavioral therapy for insomnia
  Interventions: Behavioral: ONLINE ONLY
- STEPPED CARE (Experimental): Cognitive behavioral therapy for insomnia online or therapist-led or sequentially both
  Interventions: Behavioral: STEPPED CARE

INTERVENTIONS:
Behavioral: ONLINE ONLY — Access to an online cognitive behavioral therapy for insomnia
  Arms: ONLINE ONLY
Behavioral: STEPPED CARE — A two step treatment that starts with either an online or therapist led cognitive behavioral therapy for insomnia, depending on a decision algorithm (checklist). Those with insufficient progress to the online treatment after 8 weeks are switched to a therapist-led treatment
  Arms: STEPPED CARE

SUMMARY:
This project aims to compare the effectiveness and implementation potential of two primary care friendly approaches to delivering an effective non-pharmacological intervention - cognitive behavioral therapy - for insomnia to middle aged and older adults.

DETAILED DESCRIPTION:
All participants will receive cognitive behavioral therapy for insomnia, either through an online program or through visit with a therapist specializing in behavioral sleep medicine, and is some cases both. Participants will be randomized with equal probability to an ONLINE ONLY treatment arm or to a STEPPED CARE arm, whereby they will be assigned to on line or therapist-led treatment, based on their clinical presentation; but those assigned to this arm who start treatment with an online program and do not have sufficient response after 2 months will be switched over to a therapist-led treatment.

ELIGIBILITY:
Inclusion Criteria:

* insomnia disorder

Exclusion Criteria:

* Unable to be consented in English without an interpreter
* In poor physical or mental that limits capacity to participate in study treatment (e.g., Mini-Mental State Examination score < 25)
* Unable to use the internet
* Study physician determines participation is not medically advised for any reason

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Manber, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers will share fully de-identified data on: the two primary outcomes, allocation to arm, and demographic.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available 2 years after the publication of the results pertaining to the primary aims. Data will be available for 2 years after its release
Access Criteria: Data will be shared only with investigators who have a clear and rigorous analytic plan and who sign a data use agreement with Stanford University.

REFERENCES:
- [Result] Manber R, Gumport NB, Tully IA, Kim JP, Kim B, Simpson N, Rosas LG, Zulman DM, Goldhaber-Fiebert JD, Rangel E, Dietch JR, Tutek J, Palaniappan L. Effects of a Triage Checklist to optimize insomnia treatment outcomes and reduce hypnotic use: the RCT of the effectiveness of stepped-care sleep therapy in general practice study. Sleep. 2025 Jan 13;48(1):zsae182. doi: 10.1093/sleep/zsae182. PMID 39115347
- [Derived] Tully IA, Kim JP, Simpson N, Palaniappan L, Tutek J, Gumport NB, Dietch JR, Manber R. Beliefs about prescription sleep medications and interest in reducing hypnotic use: an examination of middle-aged and older adults with insomnia disorder. J Clin Sleep Med. 2023 Jul 1;19(7):1247-1257. doi: 10.5664/jcsm.10552. PMID 36883379
- [Derived] Manber R, Tully IA, Palaniappan L, Kim JP, Simpson N, Zulman DM, Goldhaber-Fiebert JD, Rangel E, Dietch JR, Rosas LG. RCT of the effectiveness of stepped-care sleep therapy in general practice: The RESTING study protocol. Contemp Clin Trials. 2022 May;116:106749. doi: 10.1016/j.cct.2022.106749. Epub 2022 Mar 30. PMID 35367385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 388 participants signed consent. 254 were eligible and 245 were randomized to a study arm
Groups:
- ONLINE ONLY (ONLN): Online cognitive behavioral therapy for insomnia
- STEPPED CARE (STEP): Cognitive behavioral therapy for insomnia online or therapist-led or sequentially both
Period: Overall Study
Arm/Group | ONLINE ONLY (ONLN) | STEPPED CARE (STEP)
Started | 121 | 124
Triaged Checklist YES (met at least one of 5 checklist criteria) | 69 | 68
Completed | 102 | 108
Not Completed | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- ONLN: Online cognitive behavioral therapy for insomnia
- STEP: Cognitive behavioral therapy for insomnia online or therapist-led or sequentially both
- Total: Total of all reporting groups
Arm/Group | ONLN | STEP | Total
Number analyzed (Participants) | 121 | 124 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (7.90) | 62.2 (8.31) | 63.1 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 90 | 182
  Male | 29 | 34 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 12 | 19
  Not Hispanic or Latino | 108 | 110 | 218
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 21 | 22 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 88 | 89 | 177
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121 | 124 | 245
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: Score on a scale] — The ISI is an empirically validated 7-item questionnaire, with each item rated on a 4-point scale. The score is the sum of the 7 items. scores range between 0 and 28 (higher score corresponds with greater insomnia severity), with 10 as a cutoff score for identifying individuals in the community who are likely to meet criteria for insomnia disorder and 8 as a cutoff for defining remission.
  Score on a scale | 15.9 (4.25) | 15.4 (4.14) | 15.6 (4.19)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: The ISI is an empirically validated 7-item questionnaire, with each item rated on a 0 to 4 scale. The score is the sum of the 7 items. scores range between 0 and 28 (higher score corresponds with greater insomnia severity), with 10 as a cutoff score for identifying individuals in the community who are likely to meet criteria for insomnia disorder and 8 as a cutoff for defining remission.
Time Frame: at baseline and at months 2, 4, 6, 9, & 12
Population: Intent to treat sample; values for participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONLN | STEP
Number analyzed (Participants) | 121 | 124
score on a scale
  Baseline | 15.9 (4.25) | 15.4 (4.14)
  2-month: number analyzed (Participants) | 117 | 116
  2-month | 12.7 (5.00) | 11.6 (4.75)
  4-month: number analyzed (Participants) | 107 | 110
  4-month | 11.6 (4.98) | 10.0 (4.75)
  6-month: number analyzed (Participants) | 108 | 106
  6-month | 11.3 (4.93) | 9.45 (4.71)
  9-month: number analyzed (Participants) | 104 | 104
  9-month | 10.8 (4.76) | 9.12 (4.94)
  12-month: number analyzed (Participants) | 102 | 107
  12-month | 10.8 (5.16) | 8.23 (4.99)
Statistical Analysis 1: Comparison: ONLN vs STEP; Test type: Superiority; p = 0.001, Mixed Models Analysis — The a-priori threshold for statistical significance was 0.05; Mixed effects model incorporating all assessment time points; coefficient beta for change trajectory = -0.15

2. Primary Outcome: Use of Prescription Sleep Medication
Description: The average number of minimal effective doses of prescription sleep medications taken; A greater number means that the person was taking number of minimal effective doses of prescription sleep medications, with a value of 0 meaning that the person is not taking any prescription sleep medication.
Time Frame: at baseline and at months 2, 4, 6, 9, & 12
Population: Intent to treat sample; values for participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: Average number of minimal doses
Arm/Group | ONLN | STEP
Number analyzed (Participants) | 121 | 124
Average number of minimal doses
  Baseline | 0.372 (0.756) | 0.333 (0.817)
  2-month: number analyzed (Participants) | 116 | 115
  2-month | 0.357 (0.792) | 0.271 (0.660)
  4-month: number analyzed (Participants) | 107 | 110
  4-month | 0.340 (0.780) | 0.202 (0.842)
  6-month: number analyzed (Participants) | 108 | 105
  6-month | 0.352 (0.752) | 0.178 (0.638)
  9-month: number analyzed (Participants) | 104 | 102
  9-month | 0.396 (0.929) | 0.130 (0.372)
  12-month: number analyzed (Participants) | 101 | 106
  12-month | 0.375 (0.872) | 0.205 (0.874)
Statistical Analysis 1: Comparison: ONLN vs STEP; Test type: Superiority; p = 0.01, Mixed Models Analysis — The a-priori threshold for statistical significance was 0.05; Mixed effects model incorporating all assessment time points; coefficient beta for change trajectory = -0.01

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Related Impairment Questionnaire
Description: Questionnaire measuring sleep related impairment using T-scores, with a population mean of 50 and a standard deviation of 10. T-scores of 55-60 represent mild impairment; 60-70 represent moderate impairment; 70-80 represent severe impairment.
Time Frame: at baseline and at months 2, 4, 6, 9, & 12
Population: Intent to treat sample; values for participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | ONLN | STEP
Number analyzed (Participants) | 121 | 124
T score
  Baseline | 56.8 (7.48) | 56.8 (6.66)
  2-month: number analyzed (Participants) | 116 | 114
  2-month | 53.7 (7.74) | 53.4 (8.01)
  4-month: number analyzed (Participants) | 107 | 110
  4-month | 53.1 (8.25) | 52.1 (8.07)
  6-month: number analyzed (Participants) | 104 | 106
  6-month | 53.2 (7.60) | 51.0 (7.00)
  9-month: number analyzed (Participants) | 103 | 103
  9-month | 52.2 (8.45) | 50.5 (8.31)
  12-month: number analyzed (Participants) | 102 | 107
  12-month | 51.0 (8.17) | 48.2 (8.32)
Statistical Analysis 1: Comparison: ONLN vs STEP; Test type: Superiority; p = 0.0006, Mixed Models Analysis — The a-priori threshold for statistical significance was 0.05; Mixed effects model incorporating all assessment time points; coefficient beta for change trajectory = -0.24

4. Secondary Outcome: PHQ-4 (The 4 Item Patient Health Questionnaire For Anxiety and Depression)
Description: A validated questionnaire measuring depressive and anxiety symptom severity. The total score ranges between 0 and 12. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
Time Frame: at baseline and at months 2, 4, 6, 9, & 12
Population: Intent to treat sample; values for participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ONLN | STEP
Number analyzed (Participants) | 121 | 124
units on a scale
  Baseline | 2.21 (2.28) | 2.46 (2.51)
  2-month: number analyzed (Participants) | 116 | 115
  2-month | 2.63 (2.13) | 2.46 (2.51)
  4-month: number analyzed (Participants) | 108 | 110
  4-month | 2.64 (2.49) | 2.59 (2.77)
  6-month: number analyzed (Participants) | 104 | 106
  6-month | 2.51 (2.15) | 2.44 (2.23)
  9-month: number analyzed (Participants) | 103 | 103
  9-month | 2.29 (2.21) | 2.01 (1.86)
  12-month: number analyzed (Participants) | 101 | 107
  12-month | 2.34 (2.28) | 1.92 (2.12)
Statistical Analysis 1: Comparison: ONLN vs STEP; Test type: Superiority; p = 0.05, Mixed Models Analysis — The a-priori threshold for statistical significance was 0.05; Mixed effects model incorporating all assessment time points; coefficient beta for change trajectory = -0.04

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | ONLN | STEP
All-Cause Mortality (participants affected / at risk) | 1/121 | 1/124
Serious Adverse Events (participants affected / at risk) | 1/121 | 1/124
Other Adverse Events (participants affected / at risk) | 8/121 | 9/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONLN (N=121) | STEP (N=124)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Not related to study treatment
Surgical complications (Surgical and medical procedures) | 1 | 0 — Not related to study treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONLN (N=121) | STEP (N=124)
Fatigue (Psychiatric disorders) | 3 | 8
Sleepiness (Psychiatric disorders) | 5 | 8
Worsening of sleep (Psychiatric disorders) | 3 | 2
Stress about sleep (Psychiatric disorders) | 0 | 1
Discomfort due to not enough sl (Psychiatric disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03532282/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03532282/SAP_001.pdf
  • Informed Consent Form (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT03532282/ICF_002.pdf